CLINICAL TRIAL: NCT01035905
Title: Comparative Clinical Evaluation of Daily Disposable Lenses in Symptomatic Daily Disposable Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-337-C-030
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Results first posted 2010-10-19 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nelfilcon A (Experimental): Nelfilcon A contact lens
  Interventions: Device: Nelfilcon A contact lens
- Narafilcon A (Active Comparator): Narafilcon A contact lens
  Interventions: Device: Narafilcon A contact lens

INTERVENTIONS:
Device: Nelfilcon A contact lens — Daily disposable contact lens worn in a daily wear, daily disposable mode
  Arms: Nelfilcon A
Device: Narafilcon A contact lens — Daily disposable contact lens worn in a daily wear, daily disposable mode
  Arms: Narafilcon A

SUMMARY:
The purpose of this study is to evaluate the extent to which symptoms improve in symptomatic contact lens wearers when fit with one of two different daily disposable contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Currently wear daily disposable, spherical, soft lens wearers (except the two study products) for at least the past 6 months.
* Habitually wear lenses for at least 8 hours per day and 4 days per week.
* Report 2 or more qualifying symptoms with current contact lenses.
* Able to achieve visual acuity of at least 20/40 in each eye with habitual and with study lenses at dispense.
* Other protocol-defined inclusion/exclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within twelve weeks immediately prior to enrollment.
* Currently enrolled in any clinical trial.
* Any use of ocular medications, exclusive of contact lens rewetting drops.
* History of corneal or refractive surgery.
* Cylinder correction greater than 1.00 D
* Current monovision contact lens wearers.
* Other protocol-defined inclusion/exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nelfilcon A | Narafilcon A
Started | 32 | 31
Completed | 31 | 30
Not Completed | 1 | 1
Not completed — Lack of Efficacy | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nelfilcon A | Narafilcon A | Total
Number analyzed (Participants) | 32 | 31 | 63
Age Continuous [Mean (Standard Deviation); unit: years] | 31.7 (8.4) | 35.7 (11.9) | 33.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 24 | 41
  Male | 15 | 7 | 22

OUTCOME MEASURES:

1. Primary Outcome: Lens Awareness
Description: Lens awareness, as interpreted by the subject and reported by the subject in a questionnaire as a single, retrospective evaluation of 4-week's wear time. Frequency of lens awareness was measured on a 4-point scale, with 1 being never and 4 being always. Four-week ratings were compared to baseline ratings, and a negative difference (4 week minus baseline) represented an improvement.
Time Frame: 4 weeks of wear
Population: Per Protocol
Measure: Number; unit: Participants
Arm/Group | Nelfilcon A | Narafilcon A
Number analyzed (Participants) | 31 | 30
Participants | 8 | 9

ADVERSE EVENTS:
Time Frame: 63 days, duration of the study
Description: 4 weeks of exposure to product
Arm/Group | Nelfilcon A | Narafilcon A
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 0/32 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.